CLINICAL TRIAL: NCT03001544
Title: Phase 1 Single-ascending Dose-escalation Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of the Anti-alpha2-antiplasmin (α2AP) Monoclonal Antibody TS23 in Healthy Human Volunteers
Brief Title: Study of Safety and Biomarker Efficacy of TS23 in Healthy Volunteer
Acronym: TS23Phase1a
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Translational Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TS CP01-2015
Record Dates: First submitted 2016-11-11; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Thrombosis; Cerebral Ischemia; Venous Thrombosis; Pulmonary Embolism; Myocardial Infarction
MeSH Terms: conditions — Thrombosis; Brain Ischemia; Venous Thrombosis; Pulmonary Embolism; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental Ascending Dose Cohort (Experimental): TS23
  Interventions: Biological: TS23

INTERVENTIONS:
Biological: TS23 — comparison of different doses

SUMMARY:
This study is designed to determine the safety, pharmacokinetics and pharmacodynamics of a single intravenous dose of TS23 in healthy adults.

DETAILED DESCRIPTION:
This is a first-in-human, Phase 1 study of the safety, pharmacokinetics and pharmacodynamics of TS23 in healthy male volunteers.TS23 is a monoclonal antibody that inactivates alpha 2-antiplasmin. Four dose cohorts of six subjects will be studied in a single ascending dose trial at one clinical center.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Healthy males age 18 years to 60 years of age
* Body mass index ≥ 20 and ≤ 33 kg/m squared

Exclusion Criteria:

* Known allergies or hypersensitivities to blood products or derivatives or therapeutic proteins or product excipients or components of CHO cells
* Current alcohol or drug abuse or history of alcohol or drug abuse
* Participation in any trial with an investigational drug within 90 days prior to dosing
* Blood donation of more than 500 mL of blood within 90 days prior to dosing
* Any history of a bleeding or thrombotic disorder
* Any history of significant cardiac, pulmonary, renal, hepatic, neurologic, or immunologic disorder
* Over-the-counter medications, dietary supplements and herbal products (except a daily vitamin) within 14 days of drug administration or during the study
* No prescription medication for at least 14 days or 5-half-lives, whichever is longer, prior to study drug administration.
* Use of anticoagulants, fibrinolytic agents or non-steroidal anti-inflammatory medicines (except aspirin doses of 82 mg per day or less) for 2 weeks prior to and during the study
* Known hereditary fructosemia (due to sorbitol in the formulation)
* Any previous or current monoclonal antibody therapy
* History of trauma or surgery within the past 60 days or planned surgery within 30 days
* Abnormal baseline laboratory values or any laboratory values deemed clinically significant by the Investigator
* Recent history of head trauma in last 30 days prior to receiving TS23
* Unwillingness or inability to avoid contact sports or other activities with more than a small risk of head or facial trauma within 30 days of receiving TS23
* History of or risk of falls (e.g., due to dementia, frailty, etc.)
* Sexually active subjects must agree to use a reliable method of birth control (abstinence, condoms, vasectomy) and to not donate sperm for 3 months after receiving TS23

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Number and severity of adverse events post-dose | 10 weeks
  To count the number and assess the severity of treatment emergent adverse events within 10 weeks post dose

SECONDARY OUTCOMES:
Coagulation (fibrinogen, PT, aPTT) | 10 weeks
Anti-drug antibody | 16 weeks
alpha2-antiplasmin activity | 10 weeks
D-dimer | 10 weeks
Pharmacokinetic parameter, maximum concentration of TS23 | 10 weeks
  Pharmacokinetic parameter Cmax of TS23 in plasma
Pharmacokinetic parameter, half-life of TS23 | 10 weeks
  Pharmacokinetic parameter, time required for TS23 concentrations to fall by half